CLINICAL TRIAL: NCT04356716
Title: Sildenafil for Treatment of Choroidal Ischemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Donald Coleman, Professor of Clinical Ophthalmology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAM7406
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Choroidal Ischemia; Vitelliform Macular Dystrophy; Age-related Macular Degeneration; Central Serous Retinopathy; Retinitis Pigmentosa
Keywords: Sildenafil; Viagra; Revatio
MeSH Terms: conditions — Vitelliform Macular Dystrophy; Macular Degeneration; Central Serous Chorioretinopathy; Retinitis Pigmentosa | interventions — Sildenafil Citrate; Visual Acuity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the investigational sildenafil arm with a dose of 40-80mg daily, or the records review arm when taking sildenafil off-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Sildenafil (Active Comparator): Medical record review for participants that are prescribed Sildenafil off-label as part of standard of care treatment for disease.
  Interventions: Other: Standard of Care Sildenafil
- Sildenafil (Active Comparator): Participants are prescribed sildenafil 40-80 mg daily.
  Interventions: Drug: Sildenafil; Diagnostic Test: Ocular Coherence Tomography-Angiography (OCT-A); Other: Visual Acuity (VA)

INTERVENTIONS:
Drug: Sildenafil — Initial Sildenafil dosage will be weight dependent. Participants will start at 40 mg daily (20mg in the morning, 20 mg in the evening) or 60 mg daily (40mg in the morning and 20 mg in the evening). Sildenafil dosage may be increased to up to 80mg daily (20-40mg in the morning and 20-40mg in the evening) based on the response to lower doses. If the participant has not had improvement after initial treatment, the dose may be increased, at the discretion of the study physician.
  Other Names: Viagra; Revatio
  Arms: Sildenafil
Other: Standard of Care Sildenafil — Medical record review of participants that receive Sildenafil as part of standard of care.
  Other Names: Viagra; Revatio
  Arms: Standard of Care Sildenafil
Diagnostic Test: Ocular Coherence Tomography-Angiography (OCT-A) — Retinal photographs will be taken at each study visit.
  Arms: Sildenafil
Other: Visual Acuity (VA) — Visual acuity will be measured with Snellen Eye Chart at each study visit.
  Arms: Sildenafil

SUMMARY:
The hypothesis of this study is to determine if there is a benefit afforded by the use of systemic Sildenafil to patients with choroidal and retinal degenerations and dystrophies, such as vitelliform degeneration, dry and reticular age-related macular degeneration (AMD) as well as patients with hereditary and acquired retinal dystrophies such as retinitis pigmentosa and central serous retinopathy.

DETAILED DESCRIPTION:
Age-Related Macular Degeneration (AMD) is a sight-threatening visual disturbance that affects the macula in older ages. It is irreversible if the pigment epithelium is lost (dry AMD), but wet AMD can be arrested or delayed with the use of intraocular injections of one of 3 different compounds. All three drugs are injected into the eye in minute doses of usually 0.1 ml. These are usually injected at 4 to 6 week intervals and treatment may be extended for several years. Different patterns of injection times are followed but usually are monthly for 12 or more months, or monthly for 3 months and then extended observation at one to two month intervals unless vision (visual acuity) declines or Optical Coherence Tomography-angiography (OCT-A) shows recurrence of fluid or increase in size or amount of drusen (deposits of lipofuscin) in the retina. Vitelliform macular degeneration is a disorder that causes visual loss due to drusen in the macula, which have been shown to be identical to the deposits seen in macular degeneration. The goal of therapy in this proposal is to use sildenafil to increase choroidal blood flow to treat dry AMD and slow the progression of visual loss in vitelliform and age-related dry AMD as well as other macular, retinal and choroidal degenerations and dystrophies, as well as reduce or eliminate the number of injections required by slowing down transformation of dry AMD to wet AMD in treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of retinal and choroidal degenerations (reticular or vitelliform AMD or vitelliform-type subretinal drusen) or hereditary or acquired retinal dystrophies (retinitis pigmentosa or central serous retinopathy)

Exclusion Criteria:

* Diagnosis of heart disease requiring use of nitrates
* Inability to be examined monthly or bi-monthly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Jackson Coleman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Edward Harkness Eye Institute, New York, New York, United States

REFERENCES:
- [Background] Coleman DJ, Silverman RH, Rondeau MJ, Lloyd HO, Khanifar AA, Chan RV. Age-related macular degeneration: choroidal ischaemia? Br J Ophthalmol. 2013 Aug;97(8):1020-3. doi: 10.1136/bjophthalmol-2013-303143. Epub 2013 Jun 5. PMID 23740965
- [Background] Coleman DJ, Lee W, Chang S, Silverman RH, Lloyd HO, Daly S, Tsang SH. Treatment of Macular Degeneration with Sildenafil: Results of a Two-Year Trial. Ophthalmologica. 2018;240(1):45-54. doi: 10.1159/000486105. Epub 2018 Apr 25. PMID 29694963

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Record Review: Medical record review for participants that are prescribed Sildenafil off-label as part of standard of care treatment for disease.
Period: Overall Study
Arm/Group | Sildenafil | Medical Record Review
Started | 21 | 1
Completed | 21 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil | Medical Record Review | Total
Number analyzed (Participants) | 21 | 1 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 1 | 15
  >=65 years | 7 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 12
  Male | 10 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 1 | 13
  Unknown or Not Reported | 8 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 1 | 12
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 8 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 21 | 1 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Acuity (Sildenafil Group)
Description: Patients are evaluated for progression of disease/dystrophy via visual acuity (improved/stable/worsened) and appearance of fluid layer and drusen on OCT testing.
Time Frame: Up to 63 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Sildenafil
Number analyzed (Participants) | 21
logMAR
  Right eyes | 0.00 (0.21)
  Left eyes | -0.03 (0.36)

2. Primary Outcome: Change in Visual Acuity (Medical Record Review Group)
Description: as for outcome 1
Time Frame: 22 months
Measure: Number; unit: logMAR
Arm/Group | Medical Record Review
Number analyzed (Participants) | 1
logMAR
  Right eye | 0.00
  Left eye | 0.00

ADVERSE EVENTS:
Time Frame: Up to 63 months
Description: The subject in the medical review arm was not seen by research staff. No AE data was collected from this subject.
Arm/Group | Sildenafil | Medical Record Review
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/0
Other Adverse Events (participants affected / at risk) | 0/21 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04356716/Prot_SAP_000.pdf